CLINICAL TRIAL: NCT01040650
Title: Metabolic Features of Post-Myopathy Patients Associated With Statin Treatment
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left institution
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: PAM-0672
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Myopathy (Statin Associated)
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Controls: Normal Controls
- Statin associated myopathy: subjects with statin associated myopathy

SUMMARY:
Statins are a class of drugs given to lower cholesterol. Although statins are considered to be generally safe, some studies show that about 10% of people on statins develop muscle-related symptoms, from fatigue (tiredness), weakness, cramping, pain and sometimes a lifethreatening muscle breakdown condition known as rhabdomyolysis. In some, these symptoms may greatly affect their daily activities. One consideration why symptoms develop in only some patients is that they may have an underlying problem in the way their muscles use fats to produce energy. In these patients, the muscles are not able to fully utilize fats and so they become tired more easily. Fat within the muscle can also affect how your body uses a hormone called insulin, which affects your blood sugar levels. The investigators are specifically interested in previous statin users and determine if the muscle symptoms are related to changes in energy and sugar use. We propose to enroll patients who have developed muscle side effects on previous statin treatment and have since discontinued statin treatment.

Our aim is to compare the metabolic parameters in these patients to age and gender-matched normal individuals.

ELIGIBILITY:
Inclusion Criteria:

SAM Group

1. Males and females 40-65 yrs old; females must be post-menopause (>12 months since last menstrual period)
2. Developed statin-associated myopathy, defined as:

   * Documented elevated levels of CPK > 3x upper limit of normal with muscle pain, weakness, cramping during statin treatment, or
   * Diagnosed with rhabdomyolysis, or
   * Developed muscle pain, weakness, cramping during statin treatment that resulted in statin discontinuation by the subject's MD
   * Developed recurrence of muscle symptoms after resumption of statin treatment, or A score of at least 5/17 on the INQoL on screening on any of the aspects of muscle symptoms (weakness, pain, locking or tiredness) based on subject's recall at the height of the muscle symptoms
3. Able to ambulate independently (in order to perform exercise tests)
4. Muscle symptoms started/ occurred within one year of starting statin treatment or within one year of changing statin brand or dose adjustment
5. Discontinued statins at least 2 months from study inclusion date
6. 20% probability of having a cardiovascular (CV) event in the next 10 years calculated using an online CV risk calculator AND with a low or a moderate American College of Sports Medicine (ACSM) risk stratification for a cardiovascular event during a treadmill test

Normal Control Group

1. Age and gender-matched individuals who are not on statins but would otherwise be candidates for statin treatment based on ATP III guidelines and have not experienced severe muscle pain, weakness or cramping at rest or during exercise
2. Have not been diagnosed with a myopathy
3. Have no family history of a myopathy or age and gender-matched individuals who have previously been on statins and did not develop muscle side effects, and have been off statins (for other than medical reasons) for at least 2 months from study inclusion
4. 20% probability of having a cardiovascular (CV) event in the next 10 years calculated using an online CV risk calculator AND with a low or a moderate American College of Sports Medicine (ACSM) risk stratification for a cardiovascular event during a treadmill test

Exclusion Criteria:

Applies to both groups of subjects

1. Current treatment with other lipid-lowering agents, or intake of red yeast rice
2. Impaired liver or kidney function ( ALT or AST 3x upper limit of normal, creatinine 3x upper limit of normal)
3. Untreated hypo or hyperthyroidism
4. Documented history of muscle disorder or myopathy other than statin-associated myopathy or previous history of elevated CPK prior to statin exposure
5. Anemia (Hb< 110 g/dL)
6. Cancer
7. Known diabetes or fasting blood glucose >126 mg/dL
8. HIV-1 infection
9. Uncontrolled blood pressure 130/80 on two anti-hypertensive drugs
10. Currently taking beta blockers
11. Known coronary artery disease or peripheral vascular disease
12. Chronic illnesses such as lupus, rheumatoid arthritis, psoriasis
13. Long term oral, nasal, or inhaler steroid use > 6 months
14. On Hormone Therapy except for thyroid replacement
15. Alcohol consumption 40 g/day (3 glasses/day wine or beers or binge drinking 4 glasses/night)
16. Surgery in the past 6 months except for minor excision/incision procedures, 12-L electrocardiogram demonstrating old/new myocardial infarction/ ischemia or other findings that, at the investigators' discretion, may put the subject at high risk
17. Cognitive impairment that prevents comprehension of questionnaires
18. Inability to read English (questionnaire language)
19. Body mass index > 30 kg/m2
20. Physical disability or previous injury that prevents safe exercise testing
21. Not eligible for MRS (attachment)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with statin associated myopathy and normal controls
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Rockefeller University, New York, New York, United States